CLINICAL TRIAL: NCT01119573
Title: Micro RNA's Associated With Lymph Node Metastasis in Endometrial Cancer
Brief Title: Biomarkers in Tissue Samples From Patients With Stage I or Stage III Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000672415; GOG-8014
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-05

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage III endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

INTERVENTIONS:
Genetic: RNA analysis
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying at biomarkers in tissue samples from patients with stage I or stage III endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify microRNA expression patterns associated with lymph node metastasis in samples from patients with endometrial cancer.

OUTLINE: Banked tumor tissue specimens are analyzed for microRNA expression profiling by microarray analysis and reverse transcriptase-PCR assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrioid endometrial cancer

  * Stage IA, IB, IC, or IIIC disease
  * Any grade
* Enrolled and evaluated on GOG-0210 Molecular Staging Study of Endometrial Cancer

  * Consented to allow their specimens and clinical data to be collected and stored for future research
* Underwent complete surgical staging, including the following:

  * Hysterectomy
  * Bilateral oophorectomy
  * Washings as well as pelvic lymphadenectomy (sampling of four left and four right pelvic lymph nodes)
  * Para-aortic lymphadenectomy (sampling of one left and one right para-aortic lymph node)
* Sufficient high-quality frozen primary tumor for testing with ≥ 75% tumor cellularity and ≤ 10% necrosis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Association between microRNA expression and lymph node metastasis

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Principal Investigator — Simmons Cancer Center